CLINICAL TRIAL: NCT02501876
Title: Type 2 Diabetes Mellitus as Accelerator for the Progression to Alzheimer's Disease in Patients With Mild Cognitive Impairment
Brief Title: Type 2 Diabetes Mellitus as Catalyst for Alzheimer's Disease
Acronym: DIACEA
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)32/2015
Record Dates: First submitted 2015-07-16; First posted 2015-07-17 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Alzheimer´s Disease; Diabetes Mellitus Type 2
Keywords: The risk of progession; patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood will be preserved in order to perform a genetic study of 10 genes related both with type 2 diabetes and Alzheimer´s disease.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- T2D-MCI: 110 MCI subjects with type 2 diabetes. There is a retrospectiv observational study. No intervention will be performed.
  Interventions: Other: There is a retrospectiv observational study. No intervention
- nonT2D-MCI: 110 MCI subjects without diabetes. There is a retrospectiv observational study. No intervention will be performed.
  Interventions: Other: There is a retrospectiv observational study. No intervention

INTERVENTIONS:
Other: There is a retrospectiv observational study. No intervention — There is a retrospectiv observational study. No intervention will be performed

SUMMARY:
In recent years, it has been observed that the type 2 diabetic patients (DM-2) have an increased risk of developing dementia, both vascular and Alzheimer's disease (AD). The term mild cognitive impairment (MCI) describes a transition state between normal cognitive function and dementia. The annual rate of conversion to dementia in MCI patients is around 15% in the general population, regardless of the presence or absence of diabetes. At present it is not possible to identify which patients with MCI are most likely to progress to AD. On this basis, the main objective of this study is to evaluate whether the presence of diabetes and or the presence of its related genes favors the conversion of MCI to AD.

DETAILED DESCRIPTION:
In recent years, it has been observed that the type 2 diabetic patients (DM-2) have an increased risk of developing dementia, both vascular and Alzheimer's disease (AD). The term mild cognitive impairment (MCI) describes a transition state between normal cognitive function and dementia. The annual rate of conversion to dementia in MCI patients is around 15% in the general population, ie regardless of the presence or absence of diabetes. At present it is not possible to identify which patients with MCI are most likely to progress to AD. On this basis, the main objective of this study is to evaluate whether the presence of diabetes favors the conversion of MCI to AD. We propose a case-control study comparing a group of 110 diabetic patients and a group of 110 non-diabetic patients with MCI matched by age, sex and cardiovascular risk factors. The main objective is the conversion to AD between the groups and if DM-2 is an independent risk factor. The secondary objective is to investigate whether genetic mechanisms related both to AD and DM-2 are associated with the increased risk of AD in diabetic patients. We will analyze 10 genes simultaneously associated with an increased risk of diabetes and / or its complications and AD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MCI using the NBACE neuropsychological tests battery.
* Age >65 years.
* At least two years follow-up.
* 110 subjects with type 2 diabetes
* 110 subjects without diabetes
* written informed consent.

Exclusion Criteria:

* patients with cerebrovascular disease (previous stroke, intracerebral lesions, etc.), including significant vascular load according to scale Fazekas (escor˃2)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A retrospective case-control study will be conducted in the Department of Endocrinology and Nutrition Hospital Vall d'Hebron, in collaboration with the department of Neurology and Laboratory. We will review the medical records and the complete neuropsychological evaluation of 110 subjects with MCI and DM-2 matched by age, sex, and cardiovascular risk factors with 110 non-diabetic subjects with MCI. We will select the patients (diabetic or non-diabetic) with a minimum follow-up of 2 years, and whose neuropsychological assessment has been performed using the battery NBACE to ensure a uniform evaluation criteria. In addition, only patients who have determined the ApoE genotype and those who have previously undergone brain MRI will be included.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The rate of conversion to Alzheimer's disease (AD) | 6 months

SECONDARY OUTCOMES:
The presence of common alleles for Alzheimer's disease (AD) and Diabetes mellitus type 2 | 4 months
  The genetic role in the risk of conversion to AD and Diabetes mellitus type 2

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Simo Canonge, PhD, MD, Study Director — VHIR Research Institute
Locations (1):
- Vall d´Hebron University Hospital, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espinosa A, Alegret M, Valero S, Vinyes-Junque G, Hernandez I, Mauleon A, Rosende-Roca M, Ruiz A, Lopez O, Tarraga L, Boada M. A longitudinal follow-up of 550 mild cognitive impairment patients: evidence for large conversion to dementia rates and detection of major risk factors involved. J Alzheimers Dis. 2013;34(3):769-80. doi: 10.3233/JAD-122002. PMID 23271318